CLINICAL TRIAL: NCT02599155
Title: The Effect of the Hydroxyethyl Starch on Kidney Injury in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1507-061-687
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Acute Kidney Injury
Keywords: crystalloid; colloid; children; infant; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Crystalloid Solutions; Saline Solution; Colloids; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crystalloid group (Placebo Comparator): Crystalloid group receive only crystalloid for intravenous volume expansion. The same transfusion protocol is applied in both groups.
  Interventions: Drug: Crystalloid
- Colloid group (Active Comparator): Colloid group receive colloid preferentially for intravenous volume expansion, until 30 ml/kg. The same transfusion protocol is applied in both groups.
  Interventions: Drug: Colloid

INTERVENTIONS:
Drug: Crystalloid — normal saline administration for volume expansion in hypovolemic status
  Other Names: normal saline
  Arms: Crystalloid group
Drug: Colloid — HES 130/0.4 administration for volume expansion in hypovolemic status
  Other Names: HES 130/0.4
  Arms: Colloid group

SUMMARY:
The investigator will evaluate the influence of colloid administration on postoperative acute kidney injury in pediatric patients undergoing cardiac surgery under cardiopulmonary bypass.

DETAILED DESCRIPTION:
The investigator will randomly divide pediatric patients aged less than 7 years old into crystalloid and colloid groups. Crystalloid group receive only crystalloid, and colloid group receive hydroxyethyl starch (HES, 130/0.4). The maximum volume of HES is limited less than 30 ml/kg. The same transfusion protocol will be applied in both groups. From the day of operation to postoperative 7 days, glomerular filtration rate (GFR), serum creatinin level (Cr) will be checked. Acute kidney injury (AKI) is defined when there is more than 50% increase in Cr when compared to baseline level. The investigator will compare the clinical outcomes including AKI between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged less than 7 years old
* American Society of Anesthesiology (ASA) physical status 1-3

Exclusion Criteria:

* Preoperative creatinine > 1.5mg/dl
* History of dialysis
* Liver function abnormality
* Diabetes Mellitus
* History of allergic reaction
* Coagulation abnormality

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | From the day of surgery to postoperative 7 days

SECONDARY OUTCOMES:
Blood loss | From the day of surgery to postoperative 7 days
Transfusion amount | From the day of surgery to postoperative 7 days
Mechanical ventilation time | From the day of surgery to postoperative 7 days
Length of ICU stay | From the day of surgery to postoperative 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh HW, Lee JH, Kim HC, Kim EH, Song IK, Kim HS, Kim JT. The effect of 6% hydroxyethyl starch (130/0.4) on acute kidney injury in paediatric cardiac surgery: a prospective, randomised trial. Anaesthesia. 2018 Feb;73(2):205-215. doi: 10.1111/anae.14129. Epub 2017 Nov 17. PMID 29150842